CLINICAL TRIAL: NCT03563716
Title: A Phase II, Randomized, Blinded, Placebo-Controlled Study of Tiragolumab, An Anti-TIGIT Antibody, In Combination With Atezolizumab In Chemotherapy-Naïve Patients With Locally Advanced Or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Tiragolumab in Combination With Atezolizumab in Chemotherapy-Naïve Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO40290; 2018-000280-81 (EudraCT Number); 2023-508083-30-00 (EU CTIS Number)
Record Dates: First submitted 2018-04-17; First posted 2018-06-20 (Actual); Results first posted 2020-07-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Atezolizumab (Placebo Comparator): Participants will receive atezolizumab at a fixed dose of 1200 mg administered by IV infusion Q3W on Day 1 of each 21-day cycle and placebo administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Placebo
- Tiragolumab + Atezolizumab (Experimental): Participants will receive atezolizumab at a fixed dose of 1200 mg administered by intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle and tiragolumab at a dose of 600 mg administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab at a fixed dose of 1200 mg will be administered first by IV infusion Q3W on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Tiragolumab — Tiragolumab at a fixed dose of 600 mg will be administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Other Names: MTIG7192A
  Arms: Tiragolumab + Atezolizumab
Drug: Placebo — Placebo will be administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Arms: Placebo + Atezolizumab

SUMMARY:
This study will evaluate the safety and efficacy of tiragolumab plus atezolizumab compared with placebo plus atezolizumab in chemotherapy-naive patients with locally advanced unresectable or metastatic PD-L1-selected non-small cell lung cancer (NSCLC), excluding patients with a sensitizing EGFR mutation or ALK translocation.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0 or 1
* Histologically or cytologically documented locally advanced unresectable NSCLC, recurrent, or metastatic NSCLC of either squamous or non-squamous histology
* No prior systemic treatment for locally advanced unresectable or metastatic NSCLC
* Tumor PD-L1 expression
* Measurable disease, as defined by RECIST v1.1
* Life expectancy >=12 weeks
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

Cancer-Specific Exclusions:

* Patients with NSCLC known to have a sensitizing mutation in the EGFR gene or an ALK fusion oncogene
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Spinal cord compression not definitively treated with surgery and/or radiation, and/or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >=2 weeks prior to screening
* History of leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled tumor-related pain
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and/or treated with expected curative outcome

General Medical Exclusions:

* Pregnant and lactating women
* Significant cardiovascular disease
* Severe infections within 4 weeks prior to randomization
* Major surgical procedure other than for diagnosis within 4 weeks prior to randomization

Treatment-Specific Exclusions:

* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins; known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease
* Prior allogeneic bone marrow transplantation or solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Positive test for human immunodeficiency virus (HIV) and/or active hepatitis B or hepatitis C or active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2025-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (11):
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, St. Petersburg, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - Karmanos Cancer Institute, Detroit, Michigan
  - Research Medical Center, Kansas City, Missouri
  - SCRI Tennessee Oncology, Nashville, Tennessee
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
- France (5):
  - ICO Paul Papin, Angers
  - Institut Bergonié Centre Régional de Lutte Contre Le Cancer de Bordeaux Et Sud Ouest, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Hopital Nord AP-HM, Marseille
  - Institut De Cancerologie De L'Ouest, Saint-Herblain
- Serbia (3):
  - Institute of Lung Diseases Vojvodina, Kamenitz, Južnobanatski Okrug
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (10):
  - Hospital Univ Germans Trias i Pujol, Badalona, Barcelona
  - Complejo Hospitalario Universitario Insular?Materno Infantil, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Clinica Universitaria Navarra (Madrid), Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Regional Universitario de Malaga ? Hospital General, Málaga
  - Centro Medico Quironsalud Sagrado Corazon, Seville
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (5):
  - Taipei Medical University ?Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, North Dist.
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Guan X, Hu R, Choi Y, Srivats S, Nabet BY, Silva J, McGinnis L, Hendricks R, Nutsch K, Banta KL, Duong E, Dunkle A, Chang PS, Han CJ, Mittman S, Molden N, Daggumati P, Connolly W, Johnson M, Abreu DR, Cho BC, Italiano A, Gil-Bazo I, Felip E, Mellman I, Mariathasan S, Shames DS, Meng R, Chiang EY, Johnston RJ, Patil NS. Anti-TIGIT antibody improves PD-L1 blockade through myeloid and Treg cells. Nature. 2024 Mar;627(8004):646-655. doi: 10.1038/s41586-024-07121-9. Epub 2024 Feb 28. PMID 38418879
- [Derived] Cho BC, Abreu DR, Hussein M, Cobo M, Patel AJ, Secen N, Lee KH, Massuti B, Hiret S, Yang JCH, Barlesi F, Lee DH, Ares LP, Hsieh RW, Patil NS, Twomey P, Yang X, Meng R, Johnson ML. Tiragolumab plus atezolizumab versus placebo plus atezolizumab as a first-line treatment for PD-L1-selected non-small-cell lung cancer (CITYSCAPE): primary and follow-up analyses of a randomised, double-blind, phase 2 study. Lancet Oncol. 2022 Jun;23(6):781-792. doi: 10.1016/S1470-2045(22)00226-1. Epub 2022 May 13. PMID 35576957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at study sites in 6 countries.
Pre-assignment Details: Eligible patients with previously untreated, locally advanced unresectable or metastatic PD-L1-selected non-small cell lung cancer (NSCLC) were randomized 1:1 to receive either placebo plus atezolizumab or tiragolumab plus atezolizumab.
Groups:
- Placebo + Atezolizumab: Participants received atezolizumab at a fixed dose of 1200 mg administered by intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle and placebo administered by IV infusion Q3W on Day 1 of each 21-day cycle.
- Tiragolumab + Atezolizumab: Participants received atezolizumab at a fixed dose of 1200 mg administered by IV infusion Q3W on Day 1 of each 21-day cycle and tiragolumab at a dose of 600 mg administered by IV infusion Q3W on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Started | 68 | 67
Completed (Study still on-going) | 0 | 0 (One participant who died had as reason for discontinuation "Withdrawal by Subject")
Not Completed | 68 | 67
Not completed — Death | 20 | 14
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Still on Study | 45 | 50

BASELINE CHARACTERISTICS:
Groups:
- Placebo + Atezolizumab: Participants received atezolizumab at a fixed dose of 1200 mg administered by IV infusion Q3W on Day 1 of each 21-day cycle and placebo administered by IV infusion Q3W on Day 1 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.0 (9.9) | 65.8 (10.4) | 66.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 48 | 39 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 63 | 60 | 123
  Not Stated | 5 | 4 | 9
  Unknown | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 23 | 18 | 41
  White | 40 | 42 | 82
  Multiple | 1 | 0 | 1
  Unknown | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR, defined as a complete response (CR) or partial response (PR) on two consecutive occasions >/=4 weeks apart, as determined by the investigator according to RECIST v1.1. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: From baseline until a total of 80 progression free survival (PFS) events have occurred (up to approximately 11 months)
Population: Intent-to-Treat (ITT) population included all participants randomized in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 68 | 67
percentage of participants | 16.2 [6.69 to 25.66] | 31.3 [19.49 to 43.20]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratified analysis based on PD-L1 immunohistochemistry (IHC) 22C3 pharmDx, tumor histology status, and tobacco history; Test type: Superiority; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.07 to 6.14] — 95% CI for odds ratio was constructed using the Wald method

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS, defined as the time from randomization to the first occurrence of disease progression (PD), as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline).
Time Frame: From baseline until a total of 80 PFS events have occurred (up to approximately 11 months)
Population: ITT population included all participants randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 68 | 67
months | 3.58 [2.73 to 4.44] | 5.42 [4.21 to NA] — 95% Confidence Interval (CI) was not estimable as participants without documentation of progressive disease (PD) were censored.
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratified analysis based on PD-L1 IHC 22C3 pharmDx, tumor histology status, and tobacco history; Test type: Superiority; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.37 to 0.90] — Hazard ratios were estimated by Cox regression

3. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR, defined as the time from the first occurrence of a documented objective response (CR or PR) to disease progression (PD), as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline).
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Overall Survival (OS)
Description: OS, defined as the time from randomization to death from any cause.
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Serum Concentrations of Tiragolumab
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 12 Day 1 (each cycle is 21 days)
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Serum Concentrations of Atezolizumab
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 12 Day 1 (each cycle is 21 days)
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Percentage of Participants With Treatment-Emergent Anti-Drug Antibodies (ADAs)
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 12 Day 1 (each cycle is 21 days)
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: Up to primary completion date (approximately 11 months)
Description: The safety population included all participants who received at least one dose of study medication.
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 20/68 | 15/67
Serious Adverse Events (participants affected / at risk) | 24/68 | 23/67
Other Adverse Events (participants affected / at risk) | 58/68 | 60/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Atezolizumab (N=68) | Tiragolumab + Atezolizumab (N=67)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal haemorrhage (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5) | 5 (5)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Atezolizumab (N=68) | Tiragolumab + Atezolizumab (N=67)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 7 (7)
Hypothyroidism (Endocrine disorders) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 4 (5)
Constipation (Gastrointestinal disorders) | 9 (9) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 9 (12)
Nausea (Gastrointestinal disorders) | 7 (9) | 4 (4)
Vomiting (Gastrointestinal disorders) | 6 (7) | 4 (5)
Asthenia (General disorders) | 17 (18) | 17 (19)
Fatigue (General disorders) | 9 (9) | 15 (18)
Oedema peripheral (General disorders) | 3 (3) | 7 (10)
Pyrexia (General disorders) | 9 (12) | 8 (9)
Respiratory tract infection (Infections and infestations) | 5 (7) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (17) | 18 (22)
Alanine aminotransferase increased (Investigations) | 6 (6) | 3 (3)
Amylase increased (Investigations) | 2 (2) | 4 (9)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 5 (5)
Blood creatinine increased (Investigations) | 4 (4) | 1 (2)
Lipase increased (Investigations) | 2 (2) | 4 (7)
Weight decreased (Investigations) | 3 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 11 (11)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 5 (5) | 4 (5)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 9 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (12) | 13 (13)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 13 (14)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT03563716/Prot_SAP_000.pdf